CLINICAL TRIAL: NCT02094235
Title: A Phase 1/2 Study of E6005 in Pediatric Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6005-J081-102
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Dermatitis; Atopic; Pediatric; Adolescent; Child
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): E6005 0.2% ointment applied twice a day to eczema areas
  Interventions: Drug: E6005 0.2%
- 2 (Experimental): E6005 0.05% ointment applied twice a day to eczema areas
  Interventions: Drug: E6005 0.05%
- 3 (Placebo Comparator): Placebo ointment applied twice a day to eczema areas
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6005 0.05%
  Arms: 2
Drug: Placebo — 0.5 g placebo ointment
  Arms: 3
Drug: E6005 0.2%
  Arms: 1

SUMMARY:
This is a multicenter, double-blind, vehicle-control study of 0.05% and 0.2% E6005 ointment. Pediatric subjects with atopic dermatitis (AD) will be grouped into two; an elder group (childhood - adolescent: 7 to 15 years of age) and a younger group (children: 2 to 6 years of age) according to the sequential cohorts by confirming the safety.

ELIGIBILITY:
Inclusion Criteria

1. Pediatric out-patients diagnosed with AD aged 2 to 15 years at the time of written informed consent. Diagnosis for AD should be made in accordance with the "Guidelines for Management of Atopic Dermatitis" by the Japanese Dermatological Association.
2. Mild to moderate clinical symptoms appearing at baseline in areas where the application of study drug is possible, except the skin of face/head and non-dermal areas such as mucosa
3. Evaluable skin lesions appearing at baseline. "Evaluable skin lesion" means rash area of 25 to 100 cm2 in the trunk or extremities, in which at least one of dermal symptoms (erythema, exudate/eschar, excoriation or lichenification) must be moderate in severity.
4. Continuous use of an appropriate moisturizer for at least 14 days before baseline
5. Females of child-bearing potential must be negative for pregnancy test at baseline and are able to practice effective contraception during the study period including the follow-up period
6. Virile males and females of childbearing potential, who and whose partners consented to practice contraception throughout the study period after receiving an explanation using the informed consent form and the separately-prepared assent form
7. Patients whose legally acceptable representatives (caregivers) are able to consent in writing to participate in the study and who are able to adhere to the protocol requirements. For patients aged 12 years or older at the time of informed consent, written consent should be obtained from the patients as well as their legally acceptable representatives (caregivers). Also for patients aged below 12 years, written informed consent should be obtained whenever possible.

Exclusion Criteria

1. Use of biological products which may affect the pathological evaluation of AD within 6 months before the start of study treatment
2. Concurrent or recent use of certain topical or systemic medications or phototherapy without a sufficient washout period, except hydrocortisone butyrate preparations used in areas which are unsuitable for application of study drug at the discretion of the investigator
3. Currently has Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo contagious, psoriasis, connective tissue disorder, or Netherton's syndrome, etc, which may affect the pathological evaluation of AD
4. Any past history or present illness of serious allergy such as anaphylactic shock, anaphylactic reaction and anaphylactoid reaction, or any past history or present illness of drug allergic reaction or hypersensitivity
5. Has active infection that requires oral or intravenous administration of antibiotics, antifungal or antivirus agents at baseline
6. Currently has an advanced disease or highly abnormal laboratory test result that may affect the safety of subject or the implementation of the study
7. Difficulty in venous access for blood collection
8. Any past history or present illness of malignant tumor, lymphoma, leukemia or lymphoproliferative disorder, except non-melanoma skin carcinoma (e.g., squamous cell carcinoma and basal cell carcinoma) which was completely removed and has not recurred or metastasized for at least 5 years
9. Scheduled for surgery during the study
10. Concurrently enrolled in another clinical study or used any investigational drug or device within 30 days before the date of informed consent
11. Ineligible for participating in the study for other reasons, in the judgment of the investigator or subinvestigator

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of E6005 | Up to 21 Days
  The whole blood concentrations of E6005 and major metabolite will be evaluated at each visit
Number of participants with adverse events as a measure of the safety and tolerability of E6005 | Up to 21 Days
  The safety variables include adverse events, clinical laboratory parameters, vital signs and ECG results.

SECONDARY OUTCOMES:
Change from Baseline in severity score of targeted eczema | Baseline and Day 15
  For targeted eczema defined at baseline, intensity of 4 symptoms (erythema, infiltration/papulation, excoriation, and lichenification) will be assessed using a 5-grade scoring method (0: clear, 1: almost clear, 2: mild, 3: moderate, 4: severe) (maximal score: 16).
Change from Baseline in severity assessment by Investigator's Global Assessment (IGA) for targeted eczema and whole application sites | Baseline and Day 15
  Severity of AD dermal symptoms in targeted eczema and whole application sites wil be assessed based on a 6-grade scoring method (0: clear, 1: almost clear, 2: mild, 3: moderate, 4: severe, 5: most severe).
Change from Baseline in intensity of pruritus | Baseline and Day 15
  1) Interview-based pruritus scores: Subjects or caregivers (who must not be changed throughout the study) will assess the intensity of pruritus day and night within 3 days before the visit. 2) Investigator-assessed pruritus: The investigator will assess pruritus conditions by grading into 5 levels (0: clear, 1: almost clear, 2: mild, 3: moderate, 4: severe) based on the comprehensive judgments of interview and scratching behaviors.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Chitose-shi, Hokkaido
  - Eniwa-shi, Hokkaido
  - Sapporo, Hokkaido